CLINICAL TRIAL: NCT07162181
Title: Long-Term Safety of Pirtobrutinib in Participants From Study J2N-MC-JZNJ With Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma or Non-Hodgkin Lymphoma
Brief Title: Long-Term Safety of Pirtobrutinib in Participants With Previously Treated Types of Blood Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27295; J2N-MC-JZ02 (Other: Eli Lilly and Company); 2024-517760-29-00 (EU CTIS Number); J2N-MC-JZNY (Other: Eli Lilly and Company); J2N-MC-JZNJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-08-29; First posted 2025-09-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; B-cell Lymphoma
Keywords: Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell | interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pirtobrutinib (Experimental): Pirtobrutinib administered orally.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally.
  Other Names: Loxo-305; LY3527727

SUMMARY:
The purpose of this study is to find out more about the long-term safety of pirtobrutinib in participants with previously treated types of blood cancer. Participants must have chronic lymphocytic leukemia, small lymphocytic lymphoma, or non-Hodgkins lymphoma. The study is open to those who completed the original study - J2N-MC-JZNJ (NCT04849416) and continue to benefit from treatment. Treatment will be given every 12 weeks and this study is expected to last about 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled and active in the originator study, JZNJ. A participant is considered active in the study if they are receiving study intervention
* Agree to comply with contraception requirements. Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Are pregnant, or intend to become pregnant during the study, or within 30 days of last dose of study treatment or to breastfeed during the study or within 1 week of the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Grade 3 or Higher Treatment-emergent Adverse Events | Day 1 through 28 days after last dose or start of new anticancer therapy

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- China (6):
  - Beijing Cancer hospital, Beijing
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shanghai East Hospital, Shanghai
  - Blood Institute of the Chinese Academy of Medical science, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: http://vivli.org/